CLINICAL TRIAL: NCT02787434
Title: Addressing Prostate Cancer Information Disparities With eHealth Technology
Acronym: PCSPrep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jennifer Allen, Associate Professor, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1309011
Record Dates: First submitted 2016-05-19; First posted 2016-06-01 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Neoplasm
Keywords: African american men; prostate cancer screening; web-based decision aid; informed decision making; shared decision-making
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCSPrep decision aid (Experimental): All participants recruited to the trial will receive the decision aid. This a one-group study with a quasi-experiemental pre/post evaluation design.
  Interventions: Other: Prostate Cancer Screening Decision Aid

INTERVENTIONS:
Other: Prostate Cancer Screening Decision Aid — All patients recruited to the study will receive the PCSPrep decision aid. There is only 'study arm.' The Clinical Research Coordinator (CRC) will provide the patient with an iPad to complete the pre-test, PCSPrep and post-test. Individuals will see the survey questions on screen and will hear accompanying audio through headsets. Participants will: (1) be introduced to PCSPrep and the menu of activities/topics; (2) enter information about themselves for personal tailoring (e.g., risk factors); (3) participate in a values-clarification exercise to rate the personal importance of varied courses of action (i.e., pros/cons of PCS); (4) receive a printout with an individualized plan for discussing PCS with their primary care provider.
  Other Names: PCSPrep

SUMMARY:
This is a multicenter study that involves research on screening for prostate cancer. This study pilot tests a culturally appropriate decision aid (DA) for African American (AA) men that will empower them to take part in decision-making regarding prostate cancer screening (PCS). The Prostate Cancer Screening Preparation (PCSPrep) tool was designed with intend to be delivered in primary care settings with attention to patient/provider interaction. Funding for this study comes from the National Institute of Health/National Cancer Institute (1R21CA178296).

DETAILED DESCRIPTION:
STUDY AIMS AIM 1: Among AA men ages 45-70, estimate the impact of PCSPrep on primary outcomes: (a) knowledge; (b) confidence in ability to make informed decisions and communicate with provider; (c) consistency between values & PCS preferences.

AIM 2: Among primary care providers, to assess secondary outcomes: (a) perceptions regarding patient engagement in SDM; and (b) concordance with patient's ratings of SDM.

AIM 3: Among patients, providers and clinic staff, document the feasibility and acceptability of integrating PCSPrep into primary care practices.

RECRUITMENT & ENROLLMENT

Primary Care Providers Recruitment:

PCPs eligible to participate will be Emory Health Care practitioners who see at least 20 potentially eligible patients. These PCPs will be sent information from the Investigator Team and Clinic Director explaining the study We will use effective clinician recruitment procedures established in our prior work, including presentations at standing clinician meetings, meeting individually with providers, and being on site to answer questions. Ten PCPs who consent to participate will complete a brief survey following the visit from each of their enrolled patients, and allow these clinical encounters to be audio-recorded. See appendix B for post encounter survey for providers. As is standard in studies involving physicians, a financial incentive will be provided following completion of post-visit data collection for each patient when allowable and not in conflict with federal regulations. In the case of the VA hospital system, providers are not allowed to take financial incentives for research, so they will not receive this. Following the visit from each of their enrolled patients, providers will respond to a brief, online survey about the extent to which they involved the patient in the SDM process, and their perceptions regarding the quality of the communication about PCS. Total provider time in the study is estimated at 120 minutes (up to 15 enrolled patients x 10 minutes per post-encounter survey + 20 minutes of informed consent discussions).

Patient Recruitment and Enrollment:

The study will enroll AA men (age 45-70) who have not undergone prostate cancer screening (PCS) in the prior 3 years. Additional eligibility criteria will include: (1) self-reported AA race/ethnicity; (2) age 45-70; (3) English speaking. Exclusion criteria will include: personal history of prostate cancer (CaP), life expectancy of <10 years as determined by the primary care provider (PCP); or serious psychiatric conditions or cognitive impairment. Identification and recruitment of patients will be conducted by the Clinical Research Associate (CRA) under supervision of the investigators and in partnership with PCP's who opt to participate. Electronic medical records (EMR) and scheduling systems may be used to identify potentially eligible men who are scheduled for a non-acute, routine medical visit with a participating PCP during the enrollment period (i.e., Dr. Filson will access his EMR account and supervise all viewing by the CRA). See appendix D for Patient recruitment letter. Two weeks prior to a scheduled visit, eligible men will be mailed study information and an opt-out card informing them that they will be contacted by phone. Men who do not opt out will be called by the CRA, screened for eligibility, and provided with information about the study procedures. See appendix E for telephone recruitment script. Men interested in participating will be asked to arrive at the clinic 90 min prior to their scheduled visit to review study information with the CRA, provide informed consent, complete pre- and post-test and post-clinical encounter surveys, and the PSCPrep. The day prior to their scheduled visit, the CRA will call to remind them of their appointment and the opportunity to participate in this study.

INTERVENTION ADMINISTRATION PCSPrep meets the International Patient Decision Aid Standards for high quality DAs, and adheres to best practices for culturally relevant interventions.Learning objectives for participants include to: (1) understand that there is a decision to be made; (2) identify their preferred role in decision-making; (3) obtain accurate, unbiased information about benefits, limitations and potential harms of screening; (4) understand personal risk of CaP; (5) clarify one's values as they relate to the potential screening outcomes; (6) seek input from significant others, if desired; (7) develop skills for communicating with provider; (8) elicit input from provider; and (9) develop a plan for action based on desired course of action.

PCSPrep uses an audiovisual and touch-screen format on an iPad to simplify use for individuals with limited literacy and/or computer skills. It is comprised of a series of modules on the web in which professional actors describe the decision-making process, communication with a provider, and discussion of PCS. Content is delivered by actors presented as physicians who answer call-in questions in a format modeled on a health-focused television show, based on focus group feedback. Questions and discussion are presented to normalize the idea that decisions are based on individual values and preferences.

ELIGIBILITY:
Inclusion Criteria:

* African american men,
* ages 45-70 who are able to provide informed consent to participate in the educational intervention and associated data collection activities.
* English speaking

Exclusion Criteria:

* no prior personal history of prostate cancer
* no prior prostate cancer screening with the prostate specific antigen test within preceding three years
* inability to speak English

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Decision self-efficacy | Baseline (T0) upon enrollment into study; immediately following use of decision aid (PCSPrep) approx 30 min after baseline (T1); approximately one hour later, after visiting with primary care provider (T3)
  Confidence in ones ability to gather requisite information and to make an informed decision
Prostate cancer screening knowledge | Baseline (T0) upon enrollment into study; immediately following use of decision aid (PCSPrep) approximately 30 minutes after baseline (T1)
  Knowledge regarding the potential benefits, harms and limitations of prostate cancer screening
Decisional consistency | Baseline (T0) upon enrollment into study; immediately following use of decision aid (PCSPrep) approx 30 min after baseline (T1); approximately one hour later, after visiting with primary care provider (T3)
  Consistency between decision about screening and stated values regarding the pros and cons of screening

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Allen, SCD, Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Tufts University, Medford, Massachusetts
  - Emory University Hospital, Atlanta, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Plan agreement between Tufts University, Emory University, and Dana-Farber Cancer Institute

REFERENCES:
- [Derived] Allen JD, Porteny T, Kaplan A, Ladin K, Monahan K, Berry DL. Does Shared Decision-Making for Prostate Cancer Screening Among African American Men Happen? It Depends on Who You Ask. J Racial Ethn Health Disparities. 2022 Aug;9(4):1225-1233. doi: 10.1007/s40615-021-01064-x. Epub 2021 Jun 15. PMID 34129229